CLINICAL TRIAL: NCT04028635
Title: Treating the Fear of Gaining Weight. A Randomized Controlled Clinical Trial for Patients With Anorexia Nervosa
Brief Title: Treating the Fear of Gaining Weight in Anorexia Nervosa
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated with a total of 35 patients finally enrolled, due to the Sars-Cov-2 (COVID-19) global pandemic breakout and the confinement measures considered.
Sponsor: University of Barcelona (Other)
Collaborators: Hospital Sant Joan de Deu (Other); Hospital Clinic of Barcelona (Other); Hospital San Carlos, Madrid (Other); Hospital Universitari de Bellvitge (Other); Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Jose Gutierrez Maldonado, Full Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSI2015-70389-R
Record Dates: First submitted 2019-07-16; First posted 2019-07-22 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-behavioral therapy plus VR-based body exposure (Experimental): Patients assigned to this group will receive the usual CBT from the clinical unit or the hospital where they are, and additionally, six sessions of VR-based body exposure intervention. In these weekly sessions patients will go through a body exposure intervention in which the they will own a virtual avatar with their real measurements, that will progressively increase its BMI values throughout the following exposure sessions, until a healthy BMI value is reached.
  Interventions: Behavioral: Cognitive-behavioral therapy plus VR-based body exposure
- Cognitive behavioral therapy (Active Comparator): Patients assigned to this group will receive the usual treatment from the centre in which they are recruited for the study (CBT), and will have to complete the evaluations following the same schedule as the experimental group.
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy plus VR-based body exposure — Combine usual cognitive-behavioral treatment (CBT) sessions with additional five VR-based body-exposure therapy sessions.
  Arms: Cognitive-behavioral therapy plus VR-based body exposure
Behavioral: Cognitive behavioral therapy — Usual CBT
  Arms: Cognitive behavioral therapy

SUMMARY:
The main aim of this study is to develop a virtual reality (VR) embodiment-based exposure technique to improve the treatment of anorexia nervosa (AN). A systematic and hierarchical body exposure intervention in which the patient owns a virtual avatar is proposed. At first, the virtual body matches with the real measurements of the patient, then the experimenter will progressively increase Body Mass Index (BMI) values of the virtual body during the exposure sessions until a healthy BMI value is reached (e.g. BMI score of 20). In this study a VR embodiment-based technique that combines visuo-motor and a visuo-tactile stimulation procedures is proposed in order to increase illusory feelings of ownership over the virtual body. It is hypothesised that adding a VR-based body exposure intervention to the classical cognitive behavioral therapy (CBT) will significantly reduce symptomatology in AN patients.

DETAILED DESCRIPTION:
In order to evaluate the efficacy of the addition of a VR body exposure component to the usual treatment, a randomized controlled clinical trial will be conducted. 54 patients with a primary diagnosis of anorexia nervosa and a BMI > 18.5 will be randomly assigned to the experimental group receiving VR body exposure in addition to cognitive behavioral therapy or control group, which receives cognitive behavioral therapy only. Data regarding eating disorder symptomatology and body related attention will be collected before and at the end of the intervention, as well as after six months of follow-up. In the systematic and hierarchical VR body exposure intervention, which consists of 5 weekly exposure sessions, patients will gradually be exposed to increases in the BMI of their virtual avatar. Each session starts by inducing illusory feelings of ownership over the virtual body by the means of visuo-tactile and visuo-motor stimulation. Then patients are exposed to their virtual bodies in order to achieve the habituation or extinction of the anxiety response to their body image and, consequently, reduce the fear of gaining weight. During exposure, patients will be asked to focus on different parts of the virtual body, by asking what they think and feel about them. Body ownership illusion, body-related anxiety and fear of gaining weight will be assessed within each session by means of visual analogue scales.

ELIGIBILITY:
Inclusion Criteria:

* patients with primary diagnosis of anorexia nervosa (DSM-V)
* from the age of 14 years
* with BMI <18.5

Exclusion Criteria:

* visual deficits
* epilepsy or neuroleptic medication
* psychotic disorder
* bipolar disorder
* medical complications
* pregnancy
* clinical cardiac arrhythmia

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index | from pre-assessment to post-assessment after 6 weeks
  Evaluation of change in Body Mass Index
Change in Eating Disorders Inventory-3 (EDI-3) drive for thinness (EDI-DT) scale | from pre-assessment to post-assessment after 6 weeks
  Evaluation of the change in drive for thinness, with maximum possible score of 28, where higher scores indicate higher drive for thinness
Change in Eating Disorders Inventory-3 (EDI-3) body dissatisfaction (EDI-BD) scale | from pre-assessment to post-assessment after 6 weeks
  Evaluation of the change in body dissatisfaction, with maximum possible score of 40, where higher scores indicate higher body dissatisfaction
Change in Silhouette Test for Adolescents (TSA) body distortion scores | from pre-assessment to post-assessment after 6 weeks
  Evaluation of the change in body distortion in adolescents using the TSA body distortion scores, which can range from -3 to 3, with higher values indicating higher body distortion
Change in Silhouette Test for Adolescents (TSA) body dissatisfaction scores | from pre-assessment to post-assessment after 6 weeks
  Evaluation of the change in body dissatisfaction in adolescents using the TSA body dissatisfaction scores, which can range from -3 to 3, with lower scores indicating higher body dissatisfaction
Figural Drawing Scale for Body Image Assessment (BIAS-BD) body distortion scores | from pre-assessment to post-assessment after 6 weeks
  Evaluation of the change in body distortion in adults using the BIAS-BD body distortion scores, ranging from -80 to 80, with higher scores indicating higher body distortion
Figural Drawing Scale for Body Image Assessment (BIAS-BD) body dissatisfaction scores | from pre-assessment to post-assessment after 6 weeks
  Evaluation of the change in body dissatisfaction in adults using the BIAS-BD body dissatisfaction scores, ranging from -80 to 80, with higher scores indicating higher body dissatisfaction
Change in Physical Appearance State Anxiety Scale (PASTAS) | from pre-assessment to post-assessment after 6 weeks
  Evaluation of body-related anxiety using the PASTAS, with a maximum score of 32, with higher scores indicating higher body-related anxiety
Change in Body Appreciation Scale (BAS) | from pre-assessment to post-assessment after 6 weeks
  Evaluation of the change in body appreciation using the BAS, with a scale of possible scores ranging from 13-65, where higher scores indicate higher body appreciation

SECONDARY OUTCOMES:
Change in complete fixation time of the gaze towards weight-related body parts | from pre-assessment to post-assessment after 6 weeks
  Evaluation of the attentional bias towards the body using complete fixation time (evaluated in milliseconds) of the gaze towards weight-related body parts, with higher values indicating a greater attentional bias
Change in number of fixations of the gaze towards weight-related body parts | from pre-assessment to post-assessment after 6 weeks
  Evaluation of the attentional bias towards the body using the number of fixations of the gaze towards weight-related body parts, with higher values indicating a greater attentional bias

OTHER OUTCOMES:
Body-related anxiety | Up to 40 minutes. Baseline (prior to beginning the body exposure session), every two minutes during the exposure, and at the end of the body exposure session
  Visual analogue scale from 0 to 100, with higher scores indicating higher body-related anxiety
Fear of gaining weight | Up to 40 minutes. Baseline (prior to beginning the body exposure session) and at the end of the body exposure session
  Visual analogue scale from 0 to 100, with higher scores indicating higher fear of gaining weight
Body ownership illusion | Baseline (prior to beginning the body exposure session)
  Visual analogue scale from 0 to 100, with higher scores indicating higher body ownership illusion

CONTACTS AND LOCATIONS:
Overall Officials: José Gutiérrez-Maldonado, Prof. Dr., Principal Investigator — University of Barcelona
Locations (1):
- Universitat de Barcelona, Barcelona, Spain